CLINICAL TRIAL: NCT01104467
Title: Randomised, Double-blind, Placebo-controlled, Dose-escalation Study of Desmoteplase in Japanese Patients With Acute Ischemic Stroke
Brief Title: Clinical Study of Desmoteplase in Japanese Patients With Acute Ischemic Stroke
Acronym: DIAS-J
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lundbeck Japan K. K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11764A
Record Dates: First submitted 2010-04-08; First posted 2010-04-15 (Estimated); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute Ischemic Stroke; Desmoteplase; Japan; Safety; Stroke; Tolerability
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — salivary plasminogen activator alpha 1, Desmodus rotundus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Desmoteplase 70 µg/kg (Experimental)
  Interventions: Drug: Desmoteplase
- Desmoteplase 90 µg/kg (Experimental)
  Interventions: Drug: Desmoteplase
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Desmoteplase — 1 bolus injection of desmoteplase 70 µg/kg intravenous (IV)
  Arms: Desmoteplase 70 µg/kg
Drug: Desmoteplase — 1 bolus injection of desmoteplase 90 µg/kg (IV)
  Arms: Desmoteplase 90 µg/kg
Other: Placebo — 1 bolus injection of placebo IV
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate whether desmoteplase is safe and tolerated when given to Japanese patients with acute ischemic stroke

DETAILED DESCRIPTION:
The study is a safety and tolerability study of desmoteplase in Japanese patients with acute ischemic stroke. The study will test two doses

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute ischemic stroke
* Provided Informed Consent
* Male or female
* Aged between 20 and 85 years inclusive
* Treatment within 3-9 hr after onset of stroke symptoms.
* NIHSS score of 4-24 inclusive with clinical signs of hemispheric infarction
* Must receive IMP within 60 minutes after brain imaging
* Cerebral artery occlusion or high-grade stenosis in MCA

Exclusion Criteria:

* Pre-stroke mRS score of >1
* Previously exposed to desmoteplase
* Scores >2 on NIHSS question 1a indicating coma
* History or clinical presentation of ICH, subarachnoid haemorrhage (SAH), arterio-venous malformation (AVM), moyamoya disease, cerebral neoplasm or aneurysm
* Current use of oral anticoagulants and a prolonged prothrombin time (INR >1.6)
* Treated with heparin in the previous 48 hours and has a prolonged partial thromboplastin time
* Baseline platelet count <100,000/mm3
* Baseline haematocrit of <0.25
* Baseline blood glucose <50 mg/dl or >200 mg/dl
* Uncontrolled hypertension defined by a blood pressure, systolic >185 mmHg or diastolic >110 mmHg on at least 2 separate occasions at least 10 minutes apart
* Patient has hereditary or acquired hemorrhagic diathesis
* Gastrointestinal or urinary bleeding within the past 21 days
* Arterial puncture in a non-compressible site within the previous 7 days
* Another stroke or a serious head injury in the past 6 weeks
* Major surgery or serious injury, including other sites than the head, within the preceding 14 days
* Seizure at the onset of stroke
* Acute myocardial infarction (AMI) within the previous 3 weeks
* Thrombolytic within the previous 72 hr
* Pregnant

Other inclusion and exclusion criteria may apply.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of desmoteplase doses of 70 µg/kg and 90 µg/kg in Japanese patients with acute ischemic stroke as measured by the presence of symptomatic intracranial haemorrhage (sICH) within 72 hours after IMP | 90 days

SECONDARY OUTCOMES:
To evaluate the clinical improvement at Day 90 after administration of Investigational Medicinal Product (IMP) as measured by modified Rankin Scale (mRS) | 90 days
To evaluate the clinical improvement at Day 7 and 30 after administration of IMP as measured by modified Rankin Scale (mRS) | Day 7 and Day 30
To evaluate recanalisation at 18±6 hr after administration of IMP | 18±6 hr after administration of IMP
To evaluate change in infarct size at 18±6 hr relative to pre-treatment infarct size | 18±6 hr after administration
To evaluate the pharmacokinetics (PK) and pharmacodynamics (PD) of desmoteplase | 0.5 - 9 hr
To evaluate the immunogenicity of desmoteplase | Day 7, Day 30, Day 90
To explore the predictive value of different volumes of absolute mismatch for the clinical response and other objectives | Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (19):
- Japan (19):
  - JP006, Akita
  - JP021, Fukuoka
  - JP018, Hiroshima
  - JP007, Isesaki
  - JP024, Kagoshima
  - JP011, Kawasaki
  - JP015, Kobe
  - JP022, Kumamoto
  - JP012, Nagoya
  - JP026, Nishinomiya
  - JPO17, Okayama
  - JP001, Sapporo
  - JP002, Sapporo,Hokkaido
  - JP004, Sendai
  - JP005, Shibata
  - JP014, Suita
  - JP020, Tokushima
  - JP009, Tokyo
  - JP013, Toyota

REFERENCES:
- [Derived] Mori E, Minematsu K, Nakagawara J, Hasegawa Y, Nagahiro S, Okada Y, Truelsen T, Lindsten A, Ogawa A, Yamaguchi T; DIAS-J Investigators. Safety and Tolerability of Desmoteplase Within 3 to 9 Hours After Symptoms Onset in Japanese Patients With Ischemic Stroke. Stroke. 2015 Sep;46(9):2549-54. doi: 10.1161/STROKEAHA.115.009917. Epub 2015 Aug 6. PMID 26251244
- See also: Publication: "Safety and Tolerability of Desmoteplase Within 3 to 9 Hours After Symptoms Onset in Japanese Patients With Ischemic Stroke" — http://stroke.ahajournals.org/content/46/9/2549.long